CLINICAL TRIAL: NCT03688698
Title: The Relationship Between Myocardial 18F-FDG Uptake and Right Ventricular Coupling Obtained by PET/MRI Hybrid Imaging in Patients With Pulmonary Arterial Hypertension.
Brief Title: PET/MRI in PAH Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Remigiusz Kazimierczyk, MD, PhD Student, Medical University of Bialystok
Other Study IDs: 2017/25/N/NZ5/02689
Record Dates: First submitted 2018-03-26; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH
  Interventions: Radiation: PET/MRI
- Controls
  Interventions: Radiation: PET/MRI

INTERVENTIONS:
Radiation: PET/MRI — PET/MRI scans

SUMMARY:
Aim of the study is to compare novel parameters of right ventricle (RV) function from right heart catheterization (RHC) and magnetic resonance imaging (MRI) with PET-derived RV FDG uptake.

DETAILED DESCRIPTION:
Objectives In pilot study investigators aimed to compare novel parameters of right ventricle (RV) function from right heart catheterization (RHC) and magnetic resonance imaging (MRI) with PET-derived RV FDG uptake.

Background Right ventricular (RV) function is a major determinant of survival in patients with pulmonary arterial hypertension (PAH). Hemodynamic parameters like end-systolic elastance (Ees), arterial elastance (Ea), pulmonary arterial compliance (PAC) and Ees/Ea ratio have been shown to reflect RV function and prognosis in PAH. Increased RV 18F-fluoro-2-deoxyglucose (FDG) uptake in positron emission tomography (PET) was recently associated with progressive RV dysfunction in these patients.

Methods Twenty-five stable PAH patients (49.92±15.94 years) and twelve healthy subjects (control group, 44.75±13.51 years) had simultaneous PET and MRI scans performed. FDG was used as a tracer and its uptake was presented as a standardized uptake value (SUV) for both left (LV) and right ventricle.

ELIGIBILITY:
Inclusion Criteria:

- PAH

Exclusion Criteria:

The exclusion criteria were the following: patients in IV WHO class, Eisenmenger physiology, PAH associated with prevalent systemic-to-pulmonary shunts due to moderate to large defects (according to European guidelines) [16], group II, III, IV, V of pulmonary hypertension, diabetes mellitus and contraindications to cardiac MRI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled twenty-five stable adult patients diagnosed with pulmonary arterial hypertension. A diagnosis of pre-capillary pulmonary hypertension (PH) was confirmed by right heart catheterization [mean pulmonary artery pressure (mPAP) ≥25 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg] and the use of an algorithm that included perfusion lung scan, echocardiography, respiratory function tests, and computer tomography to rule out secondary PH causes according to European guidelines [16]. The control group consisted of twelve healthy controls who were matched based on sex and age. During the baseline evaluation, we performed a physical examination, six-minute walk test, laboratory tests e.g. serum B-type natriuretic peptide (BNP), morphology and renal function parameters.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in PET/MRI parameters in PAH Patients after 2 years follow-up in case of death or clinical deterioration | 2 years
  We would like to depict most significant changes in newly approved parameters from hybrid PET/MRI imaging e.g. standardised uptake value of glucose in heart, right ventricle ejection fraction, end systolic elastance, mean pulmonary pressure. This could allow us indicate possible new prognostic factors in PAH.

SECONDARY OUTCOMES:
Need of PAH targeted therapy escalation | 2 years
  Clinical worsening of patient leading to therapy escalation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kazimierczyk R, Szumowski P, Nekolla SG, Malek LA, Blaszczak P, Hladunski M, Sobkowicz B, Mysliwiec J, Kaminski KA. The impact of specific pulmonary arterial hypertension therapy on cardiac fluorodeoxyglucose distribution in PET/MRI hybrid imaging-follow-up study. EJNMMI Res. 2023 Mar 9;13(1):20. doi: 10.1186/s13550-023-00971-w. PMID 36892707
- [Derived] Kazimierczyk R, Malek LA, Szumowski P, Nekolla SG, Blaszczak P, Jurgilewicz D, Hladunski M, Sobkowicz B, Mysliwiec J, Grzywna R, Musial WJ, Kaminski KA. Multimodal assessment of right ventricle overload-metabolic and clinical consequences in pulmonary arterial hypertension. J Cardiovasc Magn Reson. 2021 May 10;23(1):49. doi: 10.1186/s12968-021-00743-2. PMID 33966635